CLINICAL TRIAL: NCT03254966
Title: Randomized, Double-blind, Placebo-controlled, Multicenter, Phase II Study to Assess the Safety and Efficacy of SHR0302 in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: Study of SHR0302 Tablets (SHR0302) as Monotherapy in Active Rheumatoid Arthritis (RA) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0302-201
Record Dates: First submitted 2017-08-15; First posted 2017-08-21 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SHR0302 dose level 1 (Experimental)
  Interventions: Drug: SHR0302
- SHR0302 dose level 2 (Experimental)
  Interventions: Drug: SHR0302
- SHR0302 dose level 3 (Experimental)
  Interventions: Drug: SHR0302
- SHR0302 dose level 4 (Experimental)
  Interventions: Drug: SHR0302
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR0302 — Oral tablets
  Arms: SHR0302 dose level 1; SHR0302 dose level 2; SHR0302 dose level 3; SHR0302 dose level 4
Drug: Placebo — Oral tablets
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of SHR0302 tablets (SHR0302) in subjects with moderate to severe active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects who are 18 - 70 (inclusive) years of age on the day of signing informed consent
* have a diagnosis of RA meeting the 2010 ACR/EULAR criteria of RA and ACR functional class I-III
* have ≥6 swollen joints (from a 66-joint count) and ≥8 tender joints (from a 68-joint count) at Screening and at Baseline, Screening serum c-reactive protein (CRP)or hsCRP > 1.2 x upper limit of laboratory normal range (ULN),or erythrocyte sedimentation rate (ESR) > 28 mm/h
* have not used any disease modifying anti-rheumatic drug (DMARD) or have an inadequate response to one or more kinds of conditional DMARDs (methotrexate, leflunomide, Chloroquine, hydroxychloroquine, sulfasalazine, minocycline, penicillamine, auranofin or injection gold preparation, and iguratimod) due to lack of efficacy or toxicity, and have agreed to be washed out from these conditional DMARDs for a period of at least 7 t1/2s prior to randomization, with the exception of antimalarials, which must be at a stable dose for at least 12 weeks prior to randomization
* Body mass index (BMI = weight/height squared (kg/m2)) within the range of 18 to 35,

Exclusion Criteria:

* current or previous RA treatment with a jak inhibitor
* current or previous RA treatment with a biologic DMARD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-10-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving an American College of Rheumatology (ACR)20 response at Week 12 | Baseline - Week 12

SECONDARY OUTCOMES:
Percentage of subjects achieving an American College of Rheumatology (ACR)20 response at Week 24 | Baseline - Week 24
Percentage of subjects achieving an American College of Rheumatology (ACR)50 response at Week 12 | Baseline - Week 12
Percentage of subjects achieving an American College of Rheumatology (ACR)50 response at Week 24 | Baseline - Week 24
Percentage of subjects achieving an American College of Rheumatology (ACR)70 response at Week 12 | Baseline - Week 12
Percentage of subjects achieving an American College of Rheumatology (ACR)70 response at Week 24 | Baseline - Week 24
Percentage of subjects achieving DAS28-3（CRP）<2.6 at Week 12 | Baseline - Week 12
Percentage of subjects achieving DAS28-3（CRP）<2.6 at Week 24 | Baseline - Week 24
Change from baseline in the Health Assessment Questionaire (HAQ-DI) at week 12 | Baseline - Week 12
Change from baseline in the Health Assessment Questionaire (HAQ-DI) at week 24 | Baseline - Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided